CLINICAL TRIAL: NCT06230562
Title: DIAGALS: Relation Between TDP-43 et Nrf-2 in ALS: a Track to Improve Diagnosis and Prognosis of the Disease: Prospective, Bicentric, Non-randomized, Open-label Study
Brief Title: DIAGALS: Relation Between Tar DNA Binding Protein(TDP)-43 et Nrf-2 in ALS: a Track to Improve Diagnosis and Prognosis of the Disease
Acronym: DIAGALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR230136
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental)
  Interventions: Biological: Blood sample
- Control group (Active Comparator)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — The intervention is to take a blood sample every 6 months for 1 year which is not part of health routine care
  Arms: Case group
Biological: Blood sample — The intervention is to take a blood sample at baseline.
  Arms: Control group

SUMMARY:
In response to oxidative stress, cells activate the Nrf-2 pathway, which induces translation of its target genes and corresponding proteins involved in the antioxidant response. This explains the interest in the Nrf-2 pathway in the pathophysiology of Amyotrophic lateral sclerosis (ALS), supported by the results of several studies and the modulatory effect of TDP-43 on the Nrf-2 pathway. Since both TDP-43 and Nrf-2 proteins are present in the peripheral blood mononuclear cells (PBMC) of ALS patients and may be correlated with disease progression, the investigators wish to explore their relationship and their application in the clinic as potential blood biomarkers for ALS.

ELIGIBILITY:
Patients group :

Inclusion Criteria:

* Men and women ≥ 18 years old
* Person affiliated to a French social security scheme or equivalent
* ALS diagnosed according to El Escorial criteria
* Diagnosis of ALS < 6 months
* Onset of symptoms < 2 years
* Signed informed consent

Non-inclusion criteria :

* Pregnant or breast-feeding
* Treatment with oral or injectable anticoagulants, antiplatelet agents (EXCEPT aspirin at the maximum authorized dosage of 160 mg per day)
* Unbalanced diabetes
* Long-term corticosteroid therapy
* Persons deprived of their liberty by judicial or administrative decision; Persons under legal protection: guardianship or curators
* Genetic mutations associated with ALS

Control group :

Inclusion criteria:

* Male or female volunteer aged 18 or over
* Person affiliated to a French social security scheme or equivalent
* Signed informed consent

Non-inclusion criteria :

* Pregnant or breast-feeding women
* Treatment with oral or injectable anticoagulants, antiplatelet agents (except aspirin at the maximum authorized dosage of 160 mg per day)
* Unbalanced diabetes
* Long-term corticosteroid therapy
* Neurological diseases
* Patient under legal protection (safeguard of justice, curators and guardianship), or in a situation of deprivation of liberty
* Genetic mutations associated with ALS

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Presence of TDP-43 aggregates in PBMC | Evolution between baseline and 6 month
  Peripheral blood samples from ALS patients and controls will be collected at inclusion and at follow-up visits for patients.
  PBMC isolation and monocyte/lymphocyte enrichment will be performed using a Percoll gradient or magnetic bead separation.
PBMC accompanied by a protein expression profile under Nrf-2 control | Evolution between baseline and 6 month
  From blood samples, RNA will be extracted from PBMCs and expression of Nrf-2 target genes will be analyzed by flow cytometry.

SECONDARY OUTCOMES:
Provide a method for identifying TDP-43 in PBMC bly flow cytometry. | At 6 month
  From blood samples, use of antibody fragments that recognize TDP-43 in the cell cytoplasm.